CLINICAL TRIAL: NCT05702944
Title: A Pilot Study for Randomized Controlled Trial on the Effect and Safety of Omitting Preoperative Alpha-adrenergic Blockade for Normotensive Pheochromocytoma
Brief Title: The Effect and Safety of Omitting Preoperative Alpha-adrenergic Blockade for Normotensive Pheochromocytoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su-jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2209-044-1357
Record Dates: First submitted 2022-11-10; First posted 2023-01-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pheochromocytoma; Paraganglioma; Adrenalectomy; Status; Adrenergics Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Phenoxybenzamine

STUDY DESIGN:
Intervention Model Description: Patients in control group take a "phenoxybenzamine" at least 2 to 5 weeks before surgery. If blood pressure is more than 130/80 mmHg in the sitting position, the patient will take a more amount of "phenoxybenzamine". If blood pressure is less than 90 mmHg in the standing position, the patient will take a less amount of "phenoxybenzamine". In the case group, there is no drug to be taken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phenoxybenzamine before surgery (Sham Comparator): Phenoxybenzamine, an alpha receptor blocker, is taken at least 2 to 5 weeks before surgery
  Interventions: Drug: Phenoxybenzamine
- No phenoxybenzamine before surgery (Active Comparator): Phenoxybenzamine, an alpha receptor blocker, is not taken before surgery
  Interventions: Drug: Phenoxybenzamine

INTERVENTIONS:
Drug: Phenoxybenzamine — Patients in sham comparator group take a phenoxybenzamine at least 2 to 5 weeks before surgery. If blood pressure is more than 130/80 mmHg in the sitting position, the patient will take a more amount of phenoxybenzamine. If blood pressure is less than 90 mmHg in the standing position, the patient will take a less amount of phenoxybenzamine. In active comparator group, there is no drug to be taken.

SUMMARY:
Pheochromocytoma and paraganglioma (PPGL) are rare neuroendocrine tumors originating from catecholamine producing chromaffin cells in the adrenal medulla and extra-adrenal paraganglia. The overall age-standardized incidence rate is 0.18 per 100,000 person-years in Korea.

The definitive treatment of PPGL is surgical excision of tumor. However, surgery is associated with a high risk of perioperative hemodynamic instability (HI). To avoid perioperative HI in patients diagnosed with PPGL, preoperative management including routine use of alpha blockade and volume expansion has been advocated by several guidelines.

While unstable hypertension and tachycardia should be controlled in patients with PPGL, there is controversial that all patients diagnosed with PPGL should undergo preoperative pharmacological treatment, especially alpha blockade. The most important risk of preoperative alpha blockade use is perioperative hypotension.

A recent study reported that patients diagnosed with PPGL postoperatively may have no further higher risk of intraoperative hypertension than those diagnosed preoperatively despite insufficient preoperatively management of PPGL.

Therefore, it is a very important to study the relationship between HI and preoperative alpha blockade in normotensive patients diagnosed with PPGL. The aim this study is to analyze the effect and safety of omitting preoperative alpha-adrenergic blockade for normotensive pheochromocytoma through a prospective randomized controlled trial. The patients is divided into two groups. The patients in control group take a phenoxybenzamine at least 2 to 5 weeks before surgery. The patients in case group do not take a phenoxybenzamine.

Primary outcome is to evaluate the percentage of time during surgery with systolic blood pressure more than 160mmHg or average blood pressure less than 60mmHg. And secondary outcomes are to evaluate hemodynamic instability in preoperative ward and postoperative ward.

DETAILED DESCRIPTION:
Pheochromocytoma and paraganglioma (PPGL) are rare neuroendocrine tumors originating from catecholamine producing chromaffin cells in the adrenal medulla and extra-adrenal paraganglia. The overall age-standardized incidence rate is 0.18 per 100,000 person-years in Korea. The classical clinical presentations that occur due to the release of catecholamine include headache, palpitation, sweating and hypertension. Excessive catecholamine release from PPGLs can induce life-threatening complication such as myocardial infarction, heart failure, cardiomyopathy, shock, arrhythmias, and stroke. The definitive treatment of PPGL is surgical excision of tumor. However, surgery is associated with a high risk of perioperative hemodynamic instability (HI). To avoid perioperative HI in patients diagnosed with PPGL, preoperative management including routine use of alpha blockade and volume expansion has been advocated by several guidelines.

While unstable hypertension and tachycardia should be controlled in patients with PPGL, there is controversial that all patients diagnosed with PPGL should undergo preoperative pharmacological treatment, especially alpha blockade. The most important risk of preoperative alpha blockade use is perioperative hypotension. The patients with prolonged preoperative alpha blockade may require intravenous fluid and vasopressors. In the recent randomized controlled trial comparing the efficacy of two different alpha blockade, 80-92% of patients reported mild to moderate side effect on alpha blockade.

The proportion of patients who are incidentally diagnosed with PPGLs are increasing. According to the recent study, the European registry for endocrine tumors revealed that incidentaloma were present in 43.4% (239/551 patients) of pheochromocytoma patients, 11.8% (65/551 patients) of patients were diagnosed as pheochromocytoma after adrenalectomy. Patients who were diagnosed with PPGL postoperatively did not undergo proper preoperative management to prevent perioperative HI. Most of them were normotensive patients and there were no specific findings on laboratory or radiologic examination suggesting PPGLs. In addition, a recent study reported that patients diagnosed with PPGL postoperatively may have no further higher risk of intraoperative hypertension than those diagnosed preoperatively despite insufficient preoperatively management of PPGL.

Therefore, it is a very important to study the relationship between HI and preoperative alpha blockade in normotensive patients diagnosed with PPGL. The department of endocrine surgery in Seoul National University Hospital intends to analyze the effect and safety of omitting preoperative alpha-adrenergic blockade for normotensive pheochromocytoma through a prospective randomized controlled trial. The patients is divided into two groups. The patients in control group take a phenoxybenzamine at least 2 to 5 weeks before surgery. If blood pressure is more than 130/80mmHg in the sitting position, the patient will take a more amount of phenoxybenzamine. If blood pressure is less than 90mmHg in the standing position, the patients will take a less amount of phenoxybenzamine. In the case group, there is no drug to be taken.

Primary outcome is to evaluate the percentage of time during surgery with systolic blood pressure more than 160mmHg or average blood pressure less than 60mmHg. And secondary outcomes are to evaluate hemodynamic instability in preoperative ward and postoperative ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 70 years old
* Patients who consented to the study and obtained consent for the study
* Patients undergoing unilateral total adrenalectomy due to normotensive pheochromocytoma/paraganglioma with less than five times of upper limits of serum metanephrine

Exclusion Criteria:

* Patients under 18 or over 70 years old
* Pregnant women
* Patients with bilateral pheochromocytoma
* Patients suspected of malignant pheochromocytoma/paraganglioma or distant metastasis
* Patients requiring preoperative intensive care unit due to severe hemodynamic instability
* Patients with hypertension (the blood pressure measured more than two times is constantly greater than 140/90 mmHg) or already taking a antihypertensive medication
* Patients with a history of coronary artery disease
* Patients with a history of arrhythmia (atrial fibrillation, Paroxysmal supraventricular tachycardia)
* Patients with a history of cerebrovascular disease (cerebral aneurysm, cerebral infarction, cerebral hemorrhage)
* Patients judged unsuitable by the person in charge of the clinical trial

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect and safety of omitting preoperative alpha blockade during surgery | during surgery
  Percentage of time during the surgery with systolic blood pressure > 160mmHg or average blood pressure < 60mmHg

SECONDARY OUTCOMES:
The effect and safety of omitting preoperative alpha blockade during surgery | during surgery
  1. Percentage of the surgery time greater than 100 times per pulse minute
  2. Average systolic/diastolic blood pressure in millimeters of mercury and pulse in beats each minutes during surgery
  3. Types and amount of antihypertensive drugs in mg per day during surgery
  4. Types and amount of vasopressor drugs in mg per day during surgery
The effect and safety of omitting preoperative alpha blockade before surgery | 3 days, 2 days, 1 day before surgery
  1. The number of times systolic blood pressure more than 130 mmHg and diastolic blood pressure more than 80mmHg in the preoperative ward
  2. The number of times of pulse rate per minute more than 80 times in the preoperative ward
The effect and safety of omitting preoperative alpha blockade after surgery | 1 day, 2 day, 2 weeks, 3 months after surgery
  1. The number of times of average blood pressure less than 60mmHg in postoperative ward
  2. Average blood pressure in postoperative ward
  3. Types and amount of antihypertensive drugs in mg per day after surgery
  4. Types and amount of vasopressor drugs in mg per day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Su-Jin Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenstrom G, Svardsudd K. Pheochromocytoma in Sweden 1958-1981. An analysis of the National Cancer Registry Data. Acta Med Scand. 1986;220(3):225-32. PMID 3776697
- [Background] Sheps SG, Jiang NS, Klee GG. Diagnostic evaluation of pheochromocytoma. Endocrinol Metab Clin North Am. 1988 Jun;17(2):397-414. PMID 3042392
- [Background] Samaan NA, Hickey RC, Shutts PE. Diagnosis, localization, and management of pheochromocytoma. Pitfalls and follow-up in 41 patients. Cancer. 1988 Dec 1;62(11):2451-60. doi: 10.1002/1097-0142(19881201)62:113.0.co;2-q. PMID 3179962
- [Background] Lenders JW, Duh QY, Eisenhofer G, Gimenez-Roqueplo AP, Grebe SK, Murad MH, Naruse M, Pacak K, Young WF Jr; Endocrine Society. Pheochromocytoma and paraganglioma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Jun;99(6):1915-42. doi: 10.1210/jc.2014-1498. PMID 24893135
- [Background] Lenders JW, Eisenhofer G, Mannelli M, Pacak K. Phaeochromocytoma. Lancet. 2005 Aug 20-26;366(9486):665-75. doi: 10.1016/S0140-6736(05)67139-5. PMID 16112304
- [Background] Pacak K. Preoperative management of the pheochromocytoma patient. J Clin Endocrinol Metab. 2007 Nov;92(11):4069-79. doi: 10.1210/jc.2007-1720. PMID 17989126
- [Background] Chen H, Sippel RS, O'Dorisio MS, Vinik AI, Lloyd RV, Pacak K; North American Neuroendocrine Tumor Society (NANETS). The North American Neuroendocrine Tumor Society consensus guideline for the diagnosis and management of neuroendocrine tumors: pheochromocytoma, paraganglioma, and medullary thyroid cancer. Pancreas. 2010 Aug;39(6):775-83. doi: 10.1097/MPA.0b013e3181ebb4f0. PMID 20664475
- [Background] Haissaguerre M, Courel M, Caron P, Denost S, Dubessy C, Gosse P, Appavoupoulle V, Belleannee G, Jullie ML, Montero-Hadjadje M, Yon L, Corcuff JB, Fagour C, Mazerolles C, Wagner T, Nunes ML, Anouar Y, Tabarin A. Normotensive incidentally discovered pheochromocytomas display specific biochemical, cellular, and molecular characteristics. J Clin Endocrinol Metab. 2013 Nov;98(11):4346-54. doi: 10.1210/jc.2013-1844. Epub 2013 Sep 3. PMID 24001749
- [Background] Kopetschke R, Slisko M, Kilisli A, Tuschy U, Wallaschofski H, Fassnacht M, Ventz M, Beuschlein F, Reincke M, Reisch N, Quinkler M. Frequent incidental discovery of phaeochromocytoma: data from a German cohort of 201 phaeochromocytoma. Eur J Endocrinol. 2009 Aug;161(2):355-61. doi: 10.1530/EJE-09-0384. Epub 2009 Jun 4. PMID 19497985
- [Background] Noshiro T, Shimizu K, Watanabe T, Akama H, Shibukawa S, Miura W, Ito S, Miura Y. Changes in clinical features and long-term prognosis in patients with pheochromocytoma. Am J Hypertens. 2000 Jan;13(1 Pt 1):35-43. doi: 10.1016/s0895-7061(99)00139-9. PMID 10678269
- [Background] Bruynzeel H, Feelders RA, Groenland TH, van den Meiracker AH, van Eijck CH, Lange JF, de Herder WW, Kazemier G. Risk Factors for Hemodynamic Instability during Surgery for Pheochromocytoma. J Clin Endocrinol Metab. 2010 Feb;95(2):678-85. doi: 10.1210/jc.2009-1051. Epub 2009 Dec 4. PMID 19965926
- [Background] Shao Y, Chen R, Shen ZJ, Teng Y, Huang P, Rui WB, Xie X, Zhou WL. Preoperative alpha blockade for normotensive pheochromocytoma: is it necessary? J Hypertens. 2011 Dec;29(12):2429-32. doi: 10.1097/HJH.0b013e32834d24d9. PMID 22025238
- [Background] Lafont M, Fagour C, Haissaguerre M, Darancette G, Wagner T, Corcuff JB, Tabarin A. Per-operative hemodynamic instability in normotensive patients with incidentally discovered pheochromocytomas. J Clin Endocrinol Metab. 2015 Feb;100(2):417-21. doi: 10.1210/jc.2014-2998. Epub 2014 Nov 18. PMID 25405501
- [Background] Buitenwerf E, Osinga TE, Timmers HJLM, Lenders JWM, Feelders RA, Eekhoff EMW, Haak HR, Corssmit EPM, Bisschop PHLT, Valk GD, Veldman RG, Dullaart RPF, Links TP, Voogd MF, Wietasch GJKG, Kerstens MN. Efficacy of alpha-Blockers on Hemodynamic Control during Pheochromocytoma Resection: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2381-91. doi: 10.1210/clinem/dgz188. PMID 31714582
- [Background] Kim JH, Lee HC, Kim SJ, Lee KE, Jung KC. Characteristics of Intraoperative Hemodynamic Instability in Postoperatively Diagnosed Pheochromocytoma and Sympathetic Paraganglioma Patients. Front Endocrinol (Lausanne). 2022 Feb 24;13:816833. doi: 10.3389/fendo.2022.816833. eCollection 2022. PMID 35282440